CLINICAL TRIAL: NCT00887302
Title: Johnson and Johnson Ethicon Metabolomics of RYGB With Gastrostomy
Brief Title: Metabolomics of Roux-en-Y Gastric Bypass (RYGB) With Gastrostomy
Status: Completed | Type: Observational
Sponsor: East Carolina University (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: J&J Ethicon
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Type II Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be collected and banked for discovery/analyses of the hypothesized GDPF and/or GDRF in subsequent studies , which are not included in the work plan or budget for this protocol extension. The basis for this proposal is the meta analysis that compares the reversal of diabetes by different bariatric surgery procedures.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Restricted food intake without rerouting food flow cohort: Obese non-diabetic patients and diabetic patients undergoing gastric band surgery will be studied before they have surgery, 1 week after the band is adjusted to restrict food intake and again after they have lost the weight equal to that which gastric bypass patients loose 3 months after surgery (to match data we already have in the current study). All patients will be studied with an intravenous glucose tolerance test to measure insulin sensitivity and IV glucose-induced insulin secretion and a meal challenge to measure the secretion of metabolites and peptides.
  Interventions: Procedure: Gastric Band
- Response to meal when a portion of the stomach is excluded from food flow cohort: Obese-diabetic patient undergoing gastric sleeve surgery will be studied before they have surgery, 1 week after surgery and again 3-6 months after surgery (to match data we already have in the current study). The patient will be studied with an intravenous glucose tolerance test to measure insulin sensitivity and insulin secretion and a meal challenge to measure the secretion of metabolites and peptides.
  Interventions: Procedure: Gastric Sleeve
- Response to meal when a portion of the GI tract is excluded from food flow cohort: In approximately 6 patients/year our surgeons have to insert a gastrostomy tube into the bypassed stomach of gastric bypass patients. This provides a unique opportunity to see the changes in metabolites and peptides in blood in response to a meal delivered to the bypassed stomach, duodenum and proximal jejunum. Since we can not anticipate which patients will require this procedure, we cannot do tests before surgery, but we will do four tests post-operatively: (1) an IV glucose tolerance test, (2) an oral meal challenge (with Hi-cal), and (3) a meal challenge (identical to that given orally/Hi-Cal) delivered through the gastrostomy tube.
  Gastrostomy subjects will also have a 4) test, a 75 gram dextrose meal challenge.
  Interventions: Procedure: Gastrostomy Tube

INTERVENTIONS:
Procedure: Gastric Band — Places a band over the upper portion of the stomach.
  Groups: Restricted food intake without rerouting food flow cohort
Procedure: Gastric Sleeve — Stapling stomach vertically to reduce size of stomach and removal of larger curve portion of the stomach
  Groups: Response to meal when a portion of the stomach is excluded from food flow cohort
Procedure: Gastrostomy Tube — Tube is inserted into the stomach that delivers nutrition directly into the stomach.
  Groups: Response to meal when a portion of the GI tract is excluded from food flow cohort

SUMMARY:
This study is an investigation of the "metabolomics of RYGB with gastrostomy."

DETAILED DESCRIPTION:
The rapid and durable remission of type II diabetes mellitis following the gastric bypass operation challenges the current concepts about the etiology of the disease. The surgery, which excludes food from the stomach, duodenum, and proximal jejunum, is quickly followed by a durable drop in glucose and insulin levels. As a result, 4 out of 5 diabetic, morbidly obese individuals who undergo the operation return to a long-term euglycemia with a prolongation of life and a reduction of health care costs.

The investigators at East Carolina University and those at Johnson and Johnson propose to further complete the profile of the upper gut by extending their observation to three additional human models. The investigators will study patients having the gastric band procedure, the gastric sleeve procedure, and those who have a gastric bypass but have a PEG tube inserted later.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-60 years of age
* BMI of 35-65
* Willing to comply with study requirements and long term follow-up
* Capable of understanding the requirements and consequences of surgery and the study
* Is scheduled to have bariatric surgery performed
* Has a negative pregnancy test

Exclusion Criteria:

* Repeat gastric bypass procedure
* Patients who are unable to hold their insulin coverage for 48 hours prior to research visits
* Patients taking TZDs

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese caucasian females between the ages of 18-60 who have had bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2012-10-12 (Actual); Study Completion 2012-10-12 (Actual)

PRIMARY OUTCOMES:
Metabolics of RYGB with Gastrostomy - Insulin | 03/25/2009-10/12/2012
  The patient will be weighed after voiding. The weight will then be used to determine the amount of insulin to be administered during the minimal model. The following formulas will be used to calculate the insulin dosages:
  REGULAR INSULIN: body mass (kg) X 0.025 U
Metabolics of RYGB with Gastrostomy - Glucose | 03/25/2009-10/12/2012
  The patient will be weighed after voiding. The weight will then be used to determine the amount of glucose to be administered during the minimal model. The following formulas will be used to calculate the glucose dosages:
  GLUCOSE: mls of 50% solution of glucose= body mass (kg) X 0.3g X 2

CONTACTS AND LOCATIONS:
Overall Officials: Walter Pories, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University Brody School of Medicine, Greenville, North Carolina, United States